CLINICAL TRIAL: NCT00734149
Title: A Prospective Study of Bortezomib in Combination With Melphalan and Prednisone for Patients With Previously Untreated Multiple Myeloma
Brief Title: Bortezomib With Melphalan and Prednisone for Multiple Myeloma
Acronym: MVP
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Pro00008089; 6019 (Other: old IRB number)
Record Dates: First submitted 2007-12-26; First posted 2008-08-14 (Estimated); Results first posted 2013-05-31 (Estimated); Last update posted 2023-11-07 (Actual); Status verified 2016-03

CONDITIONS: Multiple Myeloma
Keywords: Multiple myeloma
MeSH Terms: conditions — Multiple Myeloma | interventions — Bortezomib; Melphalan; Prednisone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Bortezomib+Melphalan+Prednisone (Experimental): Bortezomib 1.3 mg/m2 is administered intravenously in a 3-5 second bolus on days 1, 4, 8, and 11 of a 28 day cycle. Six cycles are planned. On days when both melphalan and bortezomib are given, melphalan is given at least one hour prior to bortezomib. Melphalan 6 mg/m2 is administered orally on an empty stomach daily on days 1-7 of each cycle. Prednisone 60 mg/m2 is administered orally daily on days 1-7 of each cycle.
  Interventions: Drug: Bortezomib; Drug: Melphalan; Drug: Prednisone

INTERVENTIONS:
Drug: Bortezomib
  Other Names: Velcade
Drug: Melphalan
Drug: Prednisone

SUMMARY:
The purpose of this study is to assess the efficacy of bortezomib in combination with melphalan and prednisone to achieve complete responses for patients with previously untreated multiple myeloma compared to an historical control group. This trial will also evaluate the safety and toxicity of this regimen as well as evaluate the duration of response of this regimen.

DETAILED DESCRIPTION:
Based on the need to improve front-line therapy for patients less likely to undergo transplant, the promising recent in vitro and clinical work on melphalan and bortezomib, we propose a prospective trial with bortezomib added to standard melphalan and prednisone therapy for previously untreated patients with multiple myeloma. Bortezomib 1.3 mg/m2 will be given twice weekly for two weeks and will be added to standard melphalan and prednisone on a 4-week cycle. This three-drug combination will be compared to historical data. We have treated 2 patients with relapsed disease following >2 prior regimens including high-dose therapy with autologous stem cell support. Each patient received melphalan, prednisone, and bortezomib as described below and both had marked declines in M-protein within 2 cycles. These responses have been sustained for at least 3 months and treatment was well tolerated.

Eligible patients will have histologically confirmed Multiple Myeloma (MM) having not received prior systemic therapy given with the intent to induce remission, be adults, have life expectancy greater than 3 months, adequate performance status, organ and marrow function as described in the protocol, not be pregnant, HIV positive, or taking any investigational agents. Patients must not have history of allergic reactions to study drugs or similar compounds or have uncontrolled intercurrent illness or social situation that would limit compliance with study requirements. Patients must also have the ability to give informed consent.

Study drugs will be administered on an inpatient or outpatient basis. Bortezomib 1.3 mg/m2 is administered intravenously in a 3-5 second bolus on days 1, 4, 8, and 11 of a 28 day cycle. Six cycles are planned. On days when both melphalan and bortezomib are given, melphalan is given at least one hour prior to bortezomib. Melphalan 6 mg/m2 is administered orally on an empty stomach daily on days 1-7 of each cycle. Prednisone 60 mg/m2 is administered orally daily on days 1-7 of each cycle. Supportive care measures such as antiemetics and growth factors may be given.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically confirmed multiple myeloma, defined as at least one of the following major criteria and one minor criterion or at least three minor criteria:

Major Criteria Minor Criteria Plasmacytoma on tissue biopsy Marrow plasmacytosis 10-29% Marrow plasmacytosis ≥ 30% Monoclonal protein present, less than major criteria Monoclonal protein: Lytic bone lesions

Immunoglobulin G (IgG) > 3.5 g/dl Decrease in uninvolved immunoglobulins:

Immunoglobulin A (IgA) > 2 g/dl Immunoglobulin M (IgM) < 50 mg/dl Bence Jones ≥ 1 g/24 hr IgA < 100 mg/dl IgG < 600 mg/dl

* No prior therapy
* Life expectancy greater than 3 months
* Eastern Cooperative Oncology Group (ECOG) performance status <3 (Karnofsky >40%
* Patients must have normal organ and marrow function. Patients with severe pancytopenia due to myeloma involvement of the bone marrow and patients with renal insufficiency (creatinine > 2 mg/dl) due to myeloma will also be included.
* Ability to understand and the willingness to sign a written informed consent document.

Exclusion Criteria:

* Pregnant women
* Patients may not be receiving any other investigational agents.
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to bortezomib, melphalan, or other agents used in the study.
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
* Patients with immune deficiency are at increased risk of lethal infections when treated with marrow-suppressive therapy. Therefore, HIV-positive patients receiving combination anti-retroviral therapy are excluded from the study because of possible pharmacokinetic interactions with bortezomib or other agents administered during the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2004-07; Primary Completion 2008-02 (Actual); Study Completion 2008-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Cristina Gasparetto, MD, Principal Investigator — Duke University
Locations (1):
- Duke University Medical Center, Durham, North Carolina, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment period occurred from July 2004 to December 2007 at Duke University Medical Center.
Period: Overall Study
Arm/Group | Bortezomib+Melphalan+Prednisone
Started | 45
Completed | 44
Not Completed | 1
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Arm/Group | Bortezomib+Melphalan+Prednisone
Number analyzed (Participants) | 45
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 27
  >=65 years | 18
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19
  Male | 26

OUTCOME MEASURES:

1. Primary Outcome: Response
Description: Overall response rate equals complete response and partial response per Southwest Oncology Group Criteria. Measurable, quantifiable protein criteria must be present. Acceptable protein criteria are quantitative immunoglobulin IgG, IgA, IgD, IgE or IgM and/or urine M-component (Bence-Jones protein). If both are present, the quantitative immunoglobulin will be followed for response. Complete Remission: The absence of bone marrow or blood findings of multiple myeloma. This includes disappearance of all evidence of serum and urine M-components on electrophoresis as by immunofixation studies. There must also be no evidence of increasing anemia. Partial Remission: A 50-74% reduction in the quantitative immunoglobulin, and if present, a 50-89% reduction in the urine M-component (Bence-Jones protein). Stable/No Remission): A <50% reduction I nthe quantitative immunoglobulin, or if the patient has light-chain disease only, a <50% reduction in the urine M-component (Bence-Jones protein.
Time Frame: 6 weeks following completion of treatment
Measure: Number; unit: participants
Arm/Group | Bortezomib+Melphalan+Prednisone
Number analyzed (Participants) | 44
participants | 42

2. Secondary Outcome: Number of Patients With Any Grade or Severe Adverse Event
Description: Number of patients with any grade or severe, defined as ≥ grade 3 by Common Terminology Criteria for Adverse Events (CTCAE) v4.0, adverse events as a measure of safety
Time Frame: At any time during the study and up to 30 days after stopping the study drug
Measure: Number; unit: participants
Arm/Group | Bortezomib+Melphalan+Prednisone
Number analyzed (Participants) | 45
participants | 34

3. Secondary Outcome: Median Duration of Response
Description: Duration of response is measured from date of first confirmed response until date of disease progression.
Time Frame: up to 4 years
Measure: Median (95% Confidence Interval); unit: months
Groups:
- Bortezomib+Melphalan+Prednisone: Non-ASCT: Bortezomib 1.3 mg/m2 is administered intravenously in a 3-5 second bolus on days 1, 4, 8, and 11 of a 28 day cycle. Six cycles are planned. On days when both melphalan and bortezomib are given, melphalan is given at least one hour prior to bortezomib. Melphalan 6 mg/m2 is administered orally on an empty stomach daily on days 1-7 of each cycle. Prednisone 60 mg/m2 is administered orally daily on days 1-7 of each cycle. Patients did not proceed to autologous stem cell transplant (ASCT).
- Bortezomib+Melphalan+Prednisone: ASCT: Bortezomib 1.3 mg/m2 is administered intravenously in a 3-5 second bolus on days 1, 4, 8, and 11 of a 28 day cycle. Six cycles are planned. On days when both melphalan and bortezomib are given, melphalan is given at least one hour prior to bortezomib. Melphalan 6 mg/m2 is administered orally on an empty stomach daily on days 1-7 of each cycle. Prednisone 60 mg/m2 is administered orally daily on days 1-7 of each cycle. Patients proceeded to autologous stem cell transplant (ASCT).
Arm/Group | Bortezomib+Melphalan+Prednisone: Non-ASCT | Bortezomib+Melphalan+Prednisone: ASCT
Number analyzed (Participants) | 24 | 20
months | 19.8 [14.3 to NA] — NA = many patients were censored at the time of last assessment, and therefore upper bound was not estimable- confidence intervals are extremely wide. | 27.9 [14.6 to NA] — NA = many patients were censored at the time of last assessment, and therefore upper bound was not estimable- confidence intervals are extremely wide.

ADVERSE EVENTS:
Time Frame: From first dose of study drug to 30 days after the last dose of study drug
Description: All adverse events are reported whether or not they are considered attributable to the study treatment.
Arm/Group | Bortezomib+Melphalan+Prednisone
Serious Adverse Events (participants affected / at risk) | 6/45
Other Adverse Events (participants affected / at risk) | 30/45
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Bortezomib+Melphalan+Prednisone (N=45)
Ileus, GI (functional obstruction of bowel, i.e., neuroconstipation) (Gastrointestinal disorders) | 1 (1)
Infection with unknown ANC - Lung (pneumonia) (Infections and infestations) | 1 (1)
Neuropathy: sensory (Nervous system disorders) | 2 (2)
Seizure (Nervous system disorders) | 1 (1)
Death Not Associated with CTCAE term - Disease Progression NOS (General disorders) | 2 (2)
Secondary Malignancy - possibly related to cancer treatment (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Bortezomib+Melphalan+Prednisone (N=45)
Auditory/Ear - Other (Ear and labyrinth disorders) | 1 (1)
Haptoglobin (Investigations) | 1 (1)
Hemoglobin (Blood and lymphatic system disorders) | 7 (8)
Leukocytes (total WBC) (Investigations) | 3 (5)
Neutrophils / granulocytes (ANC / AGC) (Investigations) | 4 (4)
Platelets (Investigations) | 7 (10)
Splenic function (Blood and lymphatic system disorders) | 1 (1)
Supraventricular and nodal arrhythmia - sinus bradycardia (Cardiac disorders) | 1 (1)
Hypertension (Vascular disorders) | 1 (1)
Hypotension (Vascular disorders) | 1 (4)
Fatigue (asthenia, lethargy, malaise) (General disorders) | 13 (19)
Fever (in the absence of neutropenia, defined as ANC <1.0 x 10e9/L) (General disorders) | 7 (7)
Rigors/chills (General disorders) | 4 (4)
Weight loss (Investigations) | 1 (1)
Dermatology/Skin - Other (Skin and subcutaneous tissue disorders) | 1 (1)
Dry skin (Skin and subcutaneous tissue disorders) | 1 (1)
Injection site reaction/extravasation changes (General disorders) | 1 (1)
Rash/desquamation (Skin and subcutaneous tissue disorders) | 3 (3)
Ulceration (Skin and subcutaneous tissue disorders) | 1 (1)
Hot flashes/flushes (Vascular disorders) | 1 (1)
Anorexia (Metabolism and nutrition disorders) | 3 (4)
Constipation (Gastrointestinal disorders) | 3 (4)
Dehydration (Metabolism and nutrition disorders) | 1 (1)
Dental: periodontal disease (Gastrointestinal disorders) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 2 (2)
Dysphagia (difficulty swallowing) (Gastrointestinal disorders) | 1 (1)
Flatulence (Gastrointestinal disorders) | 1 (1)
Gastrointestinal - other (Gastrointestinal disorders) | 1 (1)
Mucositis / stomatitis (clinical exam) - Oral cavity (Gastrointestinal disorders) | 2 (4)
Nausea (Gastrointestinal disorders) | 7 (8)
Heartburn / dyspepsia (Gastrointestinal disorders) | 1 (1)
Taste Alteration (dysgeusia) (Nervous system disorders) | 2 (2)
Vomiting (Gastrointestinal disorders) | 3 (3)
Febrile neutropenia - fever of unknown origin (ANC <1.0 x 10e9/L, fever >=38.5 degrees C) (Blood and lymphatic system disorders) | 3 (3)
Infection with Grade 3 or 4 neutrophils (ANC <1.0 x 10e9/L) (Infections and infestations) | 3 (3)
Infection with Grade 3 or 4 neutrophils (ANC <1.0 x 10e9/L) - lung (pneumonia) (Infections and infestations) | 1 (1)
Infection with normal ANC or Grade 1 or 2 neutrophils (Infections and infestations) | 1 (2)
Infection with unknown ANC - Urinary tract NOS (Infections and infestations) | 1 (1)
Edema: limb (General disorders) | 2 (2)
Edema: other (General disorders) | 1 (1)
ALT, SGPT (serum glutamic pyruvic transaminase) (Investigations) | 1 (1)
AST, SGOT (serum glutamic oxaloacetic transaminase) (Investigations) | 1 (1)
Potassium, serum-low (hypokalemia) (Metabolism and nutrition disorders) | 1 (1)
Sodium, serum-low (hyponatremia) (Metabolism and nutrition disorders) | 1 (1)
Fracture (Injury, poisoning and procedural complications) | 1 (1)
Joint-function (Musculoskeletal and connective tissue disorders) | 1 (1)
Mood Alteration - Anxiety (Psychiatric disorders) | 1 (1)
Mood Alteration - Depression (Psychiatric disorders) | 1 (1)
Other (General disorders) | 3 (4)
Pain - abdomen not otherwise specified (Gastrointestinal disorders) | 1 (1)
Pain - back (Musculoskeletal and connective tissue disorders) | 5 (8)
Pain - Chest / thorax not otherwise specified (General disorders) | 1 (1)
Pain - extremity - limb (Musculoskeletal and connective tissue disorders) | 1 (1)
Pain - head/headache (Nervous system disorders) | 2 (2)
Pain - other (General disorders) | 3 (4)
Cough (Respiratory, thoracic and mediastinal disorders) | 5 (8)
Dyspnea (shortness of breath) (Respiratory, thoracic and mediastinal disorders) | 7 (10)
Pneumonitis / pulmonary infiltrates (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pulmonary/upper respiratory - other (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Renal failure (Renal and urinary disorders) | 1 (1)
Urinary frequency / urgency (Renal and urinary disorders) | 3 (3)
Erectile dysfunction (Reproductive system and breast disorders) | 1 (1)
Thrombosis / thrombus / embolism (Vascular disorders) | 1 (1)
Proteinuria (Renal and urinary disorders) | 1 (1)
Neuropathy: sensory (Nervous system disorders) | 13 (17)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes